CLINICAL TRIAL: NCT05489432
Title: PREhabilitation of CAndidates for REnal Transplantation: a Hybrid Study
Brief Title: PREhabilitation of Candidates for REnal Transplantation
Acronym: PreCareTx
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Coby Annema (J.H.), PhD, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10812
Record Dates: First submitted 2022-07-28; First posted 2022-08-05 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-05

CONDITIONS: Prehabilitation; Kidney Transplant Candidates; Frailty
MeSH Terms: conditions — Frailty | interventions — Exercise; Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: An effectiveness-implementation hybrid type 1 study design comprised of a randomized controlled trial to test the effectiveness of prehabilitation to improve the overall health status of KTCs, and a mixed-methods study to gather information on its potential for further implementation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- prehabilitation group (Experimental): care as usual and pre habilitation intervention
  Interventions: Behavioral: Exercise
- control group (No Intervention): care as usual

INTERVENTIONS:
Behavioral: Exercise — A twelve-week prehabilitation program consisting of physical exercises, nutritional measures and psychosocial interventions based on the KTCs personal needs as indicated by an assessment consisting of questionnaires and physical tests. The prehabilitation program will be followed by a twelve-week consolidation program, in which the intensity and frequency of the interventions will be lower, in order to enhance the incorporation of the interventions into the daily life of the KTC. During the intervention period, participants will receive counseling by a lifestyle coach.
  Other Names: nutritional measures; stress reduction
  Arms: prehabilitation group

SUMMARY:
In this study a personalized, multi modal prehabilitation intervention will be offered to n = 64 patients on the kidney transplant waiting-list. The control group (n = 64) will receive care as usual. Based on a screening, comprised of questionnaires and physical test, eligible kidney transplant candidates who have modifiable problems on the domains of physical capacity, nutritional status or psychological well-being, will be randomly assigned to either the intervention or control group. The intervention will consist of a 12-week prehabilitation program followed by a 12 week consolidation program. Primary outcome will be frailty status as an indicator of overall health status and will be measured at screening (T0), 13 weeks (T1) and 26 weeks (T2)

DETAILED DESCRIPTION:
Rationale: The health status of kidney transplant candidates (KTCs) is often compromised due to their chronic kidney disease, comorbidities and/or dialysis. To be able to handle the stress of the upcoming transplant surgery and enhance post-operative recovery, it is important for KTCs to be in an optimal physical and psychological condition. Prehabilitation, the enhancement of a person's functional capacity in order to improve the ability to withstand a future stressor, may be an effective intervention to improve the overall health status of KTCs. Although research investigating prehabilitation in transplant populations is limited, studies showed that prehabilitation during the waiting-list period is safe and feasible, and may have a positive effect on pre- and postoperative outcomes. We hypothesized that, compared to usual care, a prehabilitation program tailored to individual patients' needs will improve the overall health status of KTCs.

Objective: To examine the effect of a multi-modal prehabilitation program on frailty and other indicators of physical and psychological fitness of KTCs during the waiting-list period and its optimal implementation in a real-world situation.

Study design: An effectiveness-implementation hybrid type 1 study design comprised of a randomized controlled trial to test the effectiveness of prehabilitation to improve the overall health status of KTCs, and a mixed-methods study to gather information on its potential for further implementation.

Study population: Adult patients, who are currently on the University Medical Center Groningen kidney transplant waiting-list or will be wait listed during the study period.

Intervention: A twelve-week prehabilitation program consisting of physical exercises, nutritional measures and psychosocial interventions based on the KTCs personal needs as indicated by an assessment consisting of questionnaires and physical tests. The prehabilitation program will be followed by a twelve-week consolidation program, in which the intensity and frequency of the interventions will be lower, in order to enhance the incorporation of the interventions into the daily life of the KTC. During the intervention period, participants will receive counseling by a lifestyle coach.

Main study parameters/endpoints: Frailty will serve as a proxy for overall health status. Therefore, the primary endpoint of this study is change in frailty status as measured by the Tilburg Frailty Indicator. Secondary endpoints include changes in physical fitness, nutritional status, psychological well-being and quality of life. Endpoints will be measured at T0 (baseline assessment), T1 (13 weeks after T0) and T2 (26 weeks after T0).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The burden for all participants (intervention and control group) will consist of filling out questionnaires (T0, 60 minutes), T1 (30 minutes) and T2 (30 minutes), completing at all three measurement points a food diary (45 minutes per measurement), to wear an activity tracker for three days, and three study visits at the UMCG in which physical tests will be performed (50-60 minutes per measurement). In total this will take ≈7 hours of their time during the 26 weeks of the study. In addition, participants in the intervention group will be asked to exercise ≈30 minutes a day and will have a weekly 10-to-15-minute counselling session by (video)call with the lifestyle coach. Efforts will differ per patient as the prehabilitation program will be tailor-made. Although the risk that patients may get injured during exercise is negligible, this will be monitored weekly by the lifestyle coach. We believe it is justified to perform the proposed study given the scarcity of data on the effectiveness of prehabilitation in KTCs and the potential of major improvements in physical functioning and psychological well-being and transplantation outcomes in this vulnerable patient group.

ELIGIBILITY:
Inclusion Criteria:

1. Adult kidney transplant candidates (≥18 years)
2. Listed for kidney transplantation on the UMCG kidney transplant waiting list at the start of the study or wait listed during the inclusion period (October 2022 - March 2025).

Exclusion Criteria:

1. Inability to read and/or speak Dutch
2. Combined organ transplantation (e.g., kidney+pancreas, kidney+liver)
3. In case of living donor kidney transplant: a transplantation planned within 3 months
4. Involved in a lifestyle intervention program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in frailty status | Baseline-week 13
  Frailty will be measured with the Tilburg Frailty Index, which measures the physical, psychological and social domain of frailty with 15 items. The total score ranges from 0-15, in which higher a score indicates a higher level of frailty
Change in frailty status | week 13- week 26
  Frailty will be measured with the Tilburg Frailty Index, which measures the physical, psychological and social domain of frailty with 15 items. The total score ranges from 0-15, in which higher a score indicates a higher level of frailty

SECONDARY OUTCOMES:
Change in functional capacity | Baseline-week 13
  The Duke Activity Status Index (DASI) will be used to measure functional capacity. The DASI consists of 12 items regarding different aspects of functioning which are answered dichotomously (yes/no). Based on the results, a total DASI score (range 0-58.2) can be calculated. A score ≤34 is indicative of low functional capacity.
Change in functional capacity | week 13- week 26
  The Duke Activity Status Index (DASI) will be used to measure functional capacity. The DASI consists of 12 items regarding different aspects of functioning which are answered dichotomously (yes/no). Based on the results, a total DASI score (range 0-58.2) can be calculated. A score ≤34 is indicative of low functional capacity.
Change in handgrip strength | Baseline-week 13
  Hand grip strength will be assessed using the Jamar Hydraulic Hand Dynamometer (Patterson Medical JAMAR 5030J1, Warrenville, Canada). Hand grip strength will be tested three times with 30 seconds of rest in between each attempt. The dominant hand will be noted in all measurements.
Change in handgrip strength | week 13- week 26
  Hand grip strength will be assessed using the Jamar Hydraulic Hand Dynamometer (Patterson Medical JAMAR 5030J1, Warrenville, Canada). Hand grip strength will be tested three times with 30 seconds of rest in between each attempt. The dominant hand will be noted in all measurements.
Change in Fat Free Mass | Baseline-week 13
  Regarding nutritional status change in fat free mass will be the main outcomes measure. Bio-impedance analysis will be performed to assess body composition. A lower percentage of fat free mass is indicative of a better nutritional status.
Change in Fat Free Mass | week 13- week 26
  Regarding nutritional status change in fat free mass will be the main outcomes measure. Bio-impedance analysis will be performed to assess body composition. A lower percentage of fat free mass is indicative of a better nutritional status.
Change in Body Mass Index | Baseline-week 13
  Body mass index will be calculated as follows: weight (in kg) divided by height (m) squared (kg/m2). A score < 20 is indicative of underweight, a score > 30 is indicative of overweight.
Change in Body Mass Index | week 13- week 26
  Body mass index will be calculated as follows: weight (in kg) divided by height (m) squared (kg/m2). A score < 20 is indicative of underweight, a score > 30 is indicative of overweight.
Change in symptoms of fatigue | Baseline-week 13
  fatigue will be measured one subscale of the Checklist Individual Strength; subjective fatigue. This subscale consists of 8 statements concerning feelings of fatigue that can be answered on a 7-point Likert scale (1 = yes, totally agree - 7 = no, totally disagree) A score of ≥27 is indicative of abnormal fatigue.
Change in symptoms of fatigue | week 13- week 26
  fatigue will be measured one subscale of the Checklist Individual Strength; subjective fatigue. This subscale consists of 8 statements concerning feelings of fatigue that can be answered on a 7-point Likert scale (1 = yes, totally agree - 7 = no, totally disagree) A score of ≥27 is indicative of abnormal fatigue.
Change in symptoms of anxiety | Baseline-week 13
  Symptoms of anxiety will be measured using the short-form of the State-Trait Anxiety Inventory consisting of 6 items rated on a 4-point intensity scale (1 = not at all; 4 = very much), resulting in a total sum score between 6 and 24. Higher scores indicate more symptoms of anxiety. A cut-off score of ≥12 is used to identify clinically relevant cases.
Change in symptoms of anxiety | week 13- week 26
  Symptoms of anxiety will be measured using the short-form of the State-Trait Anxiety Inventory consisting of 6 items rated on a 4-point intensity scale (1 = not at all; 4 = very much), resulting in a total sum score between 6 and 24. Higher scores indicate more symptoms of anxiety. A cut-off score of ≥12 is used to identify clinically relevant cases.
Change in symptoms of depression | Baseline-week 13
  Symptoms of depression will be measured using the Patient Health Questionnaire-9, a self-report questionnaire used to screen for severity of depressive symptoms, consisting of nine items and are answered on a four-point Likert scale (0 = not at all, 3 = almost every day). A total score (0-27) is calculated by adding up all scores. A score of >9 is indicative of clinically relevant symptoms of depression.
Change in symptoms of depression | week 13- week 26
  Symptoms of depression will be measured using the Patient Health Questionnaire-9, a self-report questionnaire used to screen for severity of depressive symptoms, consisting of nine items and are answered on a four-point Likert scale (0 = not at all, 3 = almost every day). A total score (0-27) is calculated by adding up all scores. A score of >9 is indicative of clinically relevant symptoms of depression.
Change in Health related Quality of Life | Baseline-week 13
  To assess Health-related Quality of life (HRQoL), the Short Form-36 (SF-36) health survey will be used. It is a 36-item, self-reported questionnaire that captures participants' perceptions of their own health and wellbeing. Based on the item scores, a physical component score (PCS) and a mental component score (MCS) will be calculated. The PCS consists of items related to general health, physical health, and role limitations due to impairment of physical health and pain. The MCS consists of items related to emotional well-being, and role limitations due to emotional problems, impaired social functioning, and impaired vitality. A higher score indicates a better perceived HRQoL
Change in Health related Quality of Life | week 13- week 26
  To assess Health-related Quality of life (HRQoL), the Short Form-36 (SF-36) health survey will be used. It is a 36-item, self-reported questionnaire that captures participants' perceptions of their own health and wellbeing. Based on the item scores, a physical component score (PCS) and a mental component score (MCS) will be calculated. The PCS consists of items related to general health, physical health, and role limitations due to impairment of physical health and pain. The MCS consists of items related to emotional well-being, and role limitations due to emotional problems, impaired social functioning, and impaired vitality. A higher score indicates a better perceived HRQoL

CONTACTS AND LOCATIONS:
Overall Officials: Coby Annema, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Quint EE, Haanstra AJ, van der Veen Y, Maring H, Berger SP, Ranchor A, Bakker SJL, Finnema E, Pol RA, Annema C; PreCareTx Investigators. PREhabilitation of CAndidates for REnal Transplantation (PreCareTx) study: protocol for a hybrid type I, mixed method, randomised controlled trial. BMJ Open. 2023 Jul 27;13(7):e072805. doi: 10.1136/bmjopen-2023-072805. PMID 37500274